CLINICAL TRIAL: NCT02663505
Title: I See You Risk Your ICU Capacity - Development Of An ICU Risk Score
Brief Title: Development of an ICU Risk Score
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Timo Iden, MD, University Hospital Schleswig-Holstein
Other Study IDs: ICU Risk Score
Record Dates: First submitted 2016-01-12; First posted 2016-01-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Development of a Risk Score for ICU Admission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients receiving either elective or emergency surgery.
  Interventions: Procedure: Patients receiving the surgery planned for them

INTERVENTIONS:
Procedure: Patients receiving the surgery planned for them — For each patient the following potential influence (risk) factors are documented:
  sex, urgency of the operation, BMI, age, ASA classification, preconditions, physical fitness, Hb value.
  In phase 2 only selected influence factors will be recorded.
  No intervention will be performed apart from the surgery planned for each patient.

SUMMARY:
Intensive care units are inevitable for high risk surgery and/or high risk patients i.e. patients with severe preconditions. However, usually the capacity of these units is limited such that at times elective surgery has to be postponed if there is no ICU capacity.

The aim of this study is to investigate potential influence/risk factors important for ICU admission in a university hospital in Germany and develop a risk score. In a second phase the risk score for ICU admission will be validated.

DETAILED DESCRIPTION:
It is one of the core duties of anesthesiologists in our hospital to identify patients with high risk for a post-surgery ICU stay upon hospital admission. We do know that there are two types of factors influencing the possibility of an ICU admission: The patient centered risk e.g. severe preconditions and the surgery centered risk depending on the type of surgery with sometimes high possibility for perioperative complications i.e. bleeding, hemodynamic instability, pulmonary complications etc. However, we do not know the effect size of these factors and, equally important, how they are correlated with one another.

The aim of this study is to model the risk of an ICU stay by patient centered and surgery centered influence factors. If a good model is obtained, this can be utilized for allocating ICU capacities in an objective fashion. The study consists of two phases. In the first phase model selection is performed. In the second phase the developed model will be validated on independent data. Data will be gathered by a data collection sheet completed by the responsible anesthesiologists in all elective and emergency surgery during a specific period of time.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years receiving surgery in the time frame of data collection with ASA classification status I-IV

Exclusion Criteria:

* Patients < 18 years
* ASA classification status > IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting inclusion criteria and receiving elective or emergency surgery
Sampling Method: Probability Sample
Enrollment: 6918 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The necessity of an ICU stay | Immediately after surgery
  This is recorded by the responsible anesthesiologist after the completion of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Grünewald, MD, Study Chair — University Hospital Schleswig-Holstein, Campus Kiel, Germany
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orsini J, Blaak C, Yeh A, Fonseca X, Helm T, Butala A, Morante J. Triage of Patients Consulted for ICU Admission During Times of ICU-Bed Shortage. J Clin Med Res. 2014 Dec;6(6):463-8. doi: 10.14740/jocmr1939w. Epub 2014 Sep 9. PMID 25247021
- [Background] Lupei MI, Chipman JG, Beilman GJ, Oancea SC, Konia MR. The association between ASA status and other risk stratification models on postoperative intensive care unit outcomes. Anesth Analg. 2014 May;118(5):989-94. doi: 10.1213/ANE.0000000000000187. PMID 24781569
- [Background] Wanderer JP, Anderson-Dam J, Levine W, Bittner EA. Development and validation of an intraoperative predictive model for unplanned postoperative intensive care. Anesthesiology. 2013 Sep;119(3):516-24. doi: 10.1097/ALN.0b013e31829ce8fd. PMID 23756454